CLINICAL TRIAL: NCT07028138
Title: Effectiveness of Electrical Stimulation With Mime Therapy Versus Electrical Stimulation With Proprioceptive Neuromuscular Facilitation on Improving Facial Asymmetry and Quality of Life in Patients With Bell's Palsy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shalamar Institute of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ShalamarIHSSSAHS
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Bell Palsy
Keywords: PNF; ES
MeSH Terms: conditions — Bell Palsy | interventions — Electric Stimulation; Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: electrical stimulation with mime therapy versus electrical stimulation with proprioceptive neuromuscular facilitation on improving facial asymmetry and quality of life in patients with Bell's palsy
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- electrical stimulation with mime therapy (Other): Mime therapy will begin with manual facial massage techniques such as tapping, stroking, and hacking, aimed at improving blood circulation and stimulating muscle activity. This will be followed by breathing and relaxation exercises to reduce muscular tension. Stretching exercises will then be performed on the affected side, including sustained pressure on trigger points in the forehead, eyes, nostrils, lips, and neck for approximately two minutes. Facial movement exercises such as eyebrow raising, eye closure, frowning, snarling, smiling, and pouting will be practiced, with each movement repeated 15 times and held for 5 to 10 seconds to encourage neuromuscular re-education. Each session will last 30 minutes and will be conducted three times per week over a six-week period.
  Interventions: Other: electrical stimulation with mime therapy
- electrical stimulation with proprioceptive neuromuscular facilitation (PNF) (Other): Group B will undergo electrical stimulation followed by proprioceptive neuromuscular facilitation (PNF). The same stimulation parameters as Group A will be used. PNF techniques will include a series of resisted facial movements such as closed-mouth smiling, lip pursing, mouth angle elevation, lower lip depression, chin tightening, and wide mouth opening, each performed with resistance and held for five seconds. These will be followed by tongue exercises including forward protrusion, elevation toward the nose, and lateral movement to both sides, with each held for five seconds. Each session will last 30 minutes and follow the same frequency and duration as Group A.
  Interventions: Other: electrical stimulation with mime therapy

INTERVENTIONS:
Other: electrical stimulation with mime therapy — A total of 38 Bell's palsy patients will be randomly selected and divided into two equal groups at Shalamar Hospital.
  Group A will receive mime therapy with electrical stimulation, including facial massage, relaxation, stretching, and facial movement exercises.
  Group B will undergo electrical stimulation followed by proprioceptive neuromuscular facilitation (PNF) with resisted facial and tongue exercises.
  Each group will receive 30-minute sessions, three times per week, for six weeks.
  Outcomes will be assessed using the Facial Disability Index (FDI), Sunnybrook Facial Grading System, and SF-12 quality of life scale.
  Evaluations will be conducted at baseline, after one month, and at a 2-3 month follow-up.
  Other Names: electrical stimulation with proprioceptive neuromuscular facilitation

SUMMARY:
To compare the effect of electrical stimulation with mime therapy versus electrical stimulation with proprioceptive neuromuscular facilitation on improving facial asymmetry and quality of life in patients with Bell's palsy.

DETAILED DESCRIPTION:
5. Introduction: (Background, Preliminary Literature Review and Significance of the Study): One paragraph related to global work on the subject, one paragraph related to local (Pakistan) work and one paragraph related to institutional work with a total of 5 to 8 references. Last paragraph should indicate the importance of work and what information/gaps are missing on topic/subject and how this study will contribute to knowledge .

Bell palsy is a sudden paralysis or weakness of the facial muscles that becomes worse over 48 hours. Bell palsy is caused by damage to the facial nerve (the 7th cranial nerve) (1). Facial nerve, which regulates facial expression muscles and transmits taste sensation from the anterior two-thirds of the tongue, becomes swollen and compressed-usually secondary to reactivation of latent herpes simplex virus type 1 (HSV-1)-in the tight bony facial canal. Thus, individuals can suddenly develop drooping of one side of the face, difficulty in blinking, hyperacusis, difficulty in moving the mouth, facial motion and expression, which makes it more difficult to communicate and tends to lower an individual's quality of life (2). Mime therapy is an advanced rehabilitation method that integrates the techniques of mime with special facial exercises to improve facial symmetry, muscle control, and emotional expression of patients with facial nerve palsy. The therapy aims to isolate facial movements, decrease synkinesis (spontaneous muscle activity), and retrain natural expressions (3). Proprioceptive neuromuscular facilitation (PNF) therapy utilizes coordinated patterns of movement to strengthen muscles and enhance neuromuscular coordination. This technique restores muscle function by activating the interaction between nerves and muscles with guided exercises (4). Electrical Stimulation (ES) applies electrical currents to activate muscles or nerves for therapeutic objectives. It helps enhance muscle strength, decrease pain, and enhance healing by causing muscle contractions or stimulation of nerves using electrodes applied on the skin. It is mostly used in the treatment of Bell's palsy(5).

Worldwide, Bell's palsy affects around 11 to 40 people per 100,000 each year with a lifetime risk of 1 in 60. It is seen most commonly in adults between 15 and 60 years of age with a mild predilection for involvement on the right side. The incidence in the United States is 24.5 per 100,000 each year. In countries like Egypt, the rate increases to 107 per 100,000 (6). In Pakistan, it differs geographically. In a study conducted in Lahore, 68.3% of the cases of facial paralysis were due to Bell's palsy and had a higher incidence in females and a right-sided predominance. In colder climates, it was most common among the 11-20 and 31-40 years of age and occurred with a peak during winter months (7) (8). European research demonstrates that PNF in combination with electrical stimulation enhances facial muscle coordination and accelerates recovery (9). In Asia, mime therapy combined with electrical stimulation has been noted to increase the strength of muscles and neuromuscular control (10). Clinical trials and reviews published most recently reveal that the use of electrical stimulation combined with either mime therapy or PNF provides more advantageous results than the use of electrical stimulation alone. Direct comparisons between the combined therapies are still limited, however, and imply that more research is warranted. There is limited direct comparison of combination therapies, leaving clinicians without evidence-based guidance and often having to make decisions based on personal choice or access to resources. This may result in suboptimal results.

Bell's palsy causes facial paralysis and loss of movement and expression. While electrical stimulation (ES), mime therapy, and proprioceptive neuromuscular facilitation (PNF) are commonly employed treatments, little is known about the combinations' effectiveness. The purpose of this study is to establish whether adding ES with mime therapy or with PNF yields better outcomes in rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Bell's Palsy Subacute and acute Bell's Palsy

Exclusion Criteria:

* UMNL facial palsy patient Non-compliant patient Patient with any psychiatric issues Patients with Dental implants Patients with any Skin condition Patients with Stroke related Bell's Palsy

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-08-28 (Estimated); Primary Completion 2025-11-29 (Estimated); Study Completion 2025-12-29 (Estimated)

PRIMARY OUTCOMES:
improving facial asymmetry | 6 weeks
  Outcome measures will include the Facial Disability Index (FDI), assessing both physical and social function, and the Sunnybrook Facial Grading System, used to evaluate facial symmetry, voluntary movement, and synkinesis before and during treatment

SECONDARY OUTCOMES:
improved Quality of life (SF-12 scores) | 6 weeks
  The SF-12 is one of the most widely used instruments for assessing self-reported health-related quality of life , A score of <40 in either PCS or MCS is used as a cut-off to indicate impaired or poor quality of life.